CLINICAL TRIAL: NCT03706326
Title: Combination Therapy of Anti-MUC1 CAR T Cells and PD-1 Knockout Engineered T Cells for Advanced Esophageal Cancer
Brief Title: CAR T and PD-1 Knockout Engineered T Cells for Esophageal Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Guangdong Pharmaceutical University (Other)
Collaborators: Guangzhou Anjie Biomedical Technology Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Size Chen, Associate Professor, The First Affiliated Hospital of Guangdong Pharmaceutical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-6301
Record Dates: First submitted 2018-10-11; First posted 2018-10-16 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Advanced Esophageal Cancer
Keywords: Esophageal cancer; Neoplasms, Esophageal; Cancer of Esophagus; Solid tumor
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment with Anti-MUC1 CAR-T cells (Experimental): Anti-MUC1 CAR-T cells will be prepared ex vivo using the T cells from the patients and infused back to the patients.
  Interventions: Biological: Anti-MUC1 CAR-T cells
- Combination Therapy: CAR-T combining PD-1 knockout T Cells (Experimental): Anti-MUC1 CAR-T cells and PD-1 knockout Engineered T cells will be prepared ex vivo using the T cells from the patients and infused back to the patients.
  Interventions: Combination Product: CAR-T combined with PD-1 Knockout T cells
- Treatment with PD-1 knockout Engineered T cells (Experimental): PD-1 knockout Engineered T cells will be prepared ex vivo using the T cells from the patients and infused back to the patients.
  Interventions: Biological: PD-1 knockout Engineered T cells

INTERVENTIONS:
Biological: Anti-MUC1 CAR-T cells — Using the T cells from the patients' blood to produce anti-MUC1 CAR-T Cells and then the cells will be infused back to the patients.
  Arms: Treatment with Anti-MUC1 CAR-T cells
Biological: PD-1 knockout Engineered T cells — Using the T cells from the blood of the patients to prepare PD-1 knockout T cells, then the cells will be infused back to the patients.
  Arms: Treatment with PD-1 knockout Engineered T cells
Combination Product: CAR-T combined with PD-1 Knockout T cells — Using the T cells from the blood of the patients to prepare anti-MUC1 CAR-T Cells and PD-1 knockout T cells, then the cells will be infused back to the patients
  Arms: Combination Therapy: CAR-T combining PD-1 knockout T Cells

SUMMARY:
The study is to assess the safety and efficacy of the immunotherapies using anti-MUC1 CAR T cells and /or PD-1 knockout engineered T cells in the treatment of patients with advanced esophageal cancer.

DETAILED DESCRIPTION:
This is a combined phase 1 and 2 clinical study. The aim of the study is to assess the safety and efficacy of the immunotherapies using anti- MUC1 CAR T cells alone, anti- MUC1 CAR T combining PD-1 knockout engineered T cells, and PD-1 knockout engineered T cell only in the treatment of patients with advanced esophageal cancer. The treatment outcomes from each group will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of advanced esophageal cancer (phase IIIb-IV) according to NCCN clinical practice guidelines in Oncology:Esophageal and Esophagogastric Junction Cancers (2018.V1).
* MUC1 is highly expressed in malignancy tissues by immuno-histochemical (IHC).
* Eastern cooperative oncology group (ECOG) performance status of 0-1 or karnofsky performance status (KPS) score is higher than 60.
* Patients have a life expectancy > 12 weeks.
* Adequate venous access for apheresis or venous sampling, and no other contraindications for leukapheresis.
* Negative pregnancy test for females of child-bearing potentials.
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements: White blood cell count (WBC) ≥ 2500c/ml, Platelets ≥ 50×10^9/L, Hb ≥ 9.0g/dL, lymphocyte (LY) ≥ 0.7×10^9/L, LY% ≥ 15%, Alb ≥ 2.8g/dL, serum lipase and amylase < 1.5×upper limit of normal, serum creatinine ≤ 2.5mg/dL, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 5×upper limit of normal, serum total bilirubin ≤ 2.0mg/dL. These tests must be conducted within 7 days prior to registration.
* Signed informed consent form.

Exclusion Criteria:

* Number of T cells is less than 10% or the amplification of the T cells via artificial antigen presenting cell (aAPC) stimulation is less than 5 times.
* Patients with symptomatic central nervous system (CNS) involvement.
* Pregnant or nursing women.
* Known HIV, HBV and HCV infection.
* Serious illness or medical condition which would not permit the patient to be managed according to the protocol, including active uncontrolled infection, major cardiovascular, coagulation disorders, respiratory or immune system, myocardial infarction, cardiac arrhythmias, obstructive/restrictive pulmonary disease, or psychiatric or emotional disorders.
* History of severe immediate hypersensitivity to any of the agents including cyclophosphamide, fludarabine, or aldesleukin.
* Concurrent use of systemic steroids. Recent or current use of inhaled steroids is not exclusionary.
* Previously treatment with any gene therapy products.
* The existence of unstable or active ulcers or gastrointestinal bleeding. Patients with portal vein vascular invasion or extrahepatic, are excluded from this study.
* Patients with a history of organ transplantation or are waiting for organ transplantation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-09-28 (Actual); Primary Completion 2021-09-28 (Estimated); Study Completion 2021-09-28 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events and dose limiting toxicities as assessed by CTCAE v4.0 | approximately 12 months
  Safety and tolerability of dose of CART-cells and PD-1 Knockout T cells will be assessed using CTCAE v4.0.

SECONDARY OUTCOMES:
Response Rate | 12 months
  Will be assessed according to the revised RECIST guideline v1.1
Overall Survival - OS | Up to 24 months
  Measure the time from enrollment to death
Progression free survival - PFS | Up to 12 months
  Time from enrollment to date of first documented progression or date of death.
Median CAR-T cell persistence | 3 years
  Will be measured by quantitative RT-PCR

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - First Affiliated Hospital of Guangdong Pharmaceutical University, Guangzhou, Guangdong
  - Professor Size Chen, Guangzhou, Guangdong